CLINICAL TRIAL: NCT06870500
Title: Card14gene (rs34367357 ) Polymorphism in Egyptian Psoriatic and Psoriatic Arthritis Patient and Its Relation With Response to Methotrexate
Brief Title: Card14gene (rs34367357 ) Polymorphism in Egyptian Psoriatic and Psoriatic Arthritis Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Marwa Naguib Ahmed, Resident of Dermatology , venereology and andrology at Faculty of medicine, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Card14gene polymorphism
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): About 20 patients with psoriasis
  Interventions: Drug: Methotrexate
- Group B (Active Comparator): About 20 psoriatic arthritis
  Interventions: Drug: Methotrexate
- Group C (Placebo Comparator): About 10 healthy control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — 1. Assess the response of psoriasis and psoriatic arthritis to Methotrexate.
  2. Assess the relation between Card14 gene(rs 34367357 ) Polymorphism in psoriatic and psoriatic arthritis patients and their clinical response to methotrexate
  Other Names: Card14 gene(rs 34367357 )
  Arms: Group A; Group B
Drug: Placebo — Placebo
  Arms: Group C

SUMMARY:
Psoriasis is a chronic, immune-mediated, multisystemic, inflammatory disease caused by the interaction of multiple susceptibility genes and environmental factors that affects 1-3% of the population worldwide .Psoriasis also is a chronic inflammatory skin disease characterized by scaly indurated erythema.

Psoriatic arthritis (PsA) is an autoimmune and chronic musculoskeletal disorder that is associated with psoriasis of the skin . Its presentation can vary from subtle manifestations to highly destructive forms. Joint pain, stiffness and swelling are the most common symptoms.

DETAILED DESCRIPTION:
PsA is a complex inflammatory disease with heterogeneous clinical features, which complicates psoriasis in 30% of patients .

The exact aetiopathogenesis of psoriasis is not completely explained. Pathological mechanism involves skin inflammation and hyperproliferation of keratinocytes induced innate and adaptive immune cells. Genetic, immunological and environmental factors are considered the most important aetiologies.

Psoriasis is a chronic relapsing disease, which often necessitates a long-term therapy. Mild to moderate psoriasis can be treated topically with a combination of glucocorticoids, vitamin D analogues, and phototherapy. Moderate to severe psoriasis often requires systemic treatment. The presence of comorbidities such as psoriasis arthritis is also highly relevant in treatment selection.

Methotrexate (MTX) has remained the backbone of the treatment for moderate to severe psoriasis ever since its first use nearly half a century ago.

Over the years, its high efficacy, low cost, relative ease of administration and usefulness in concomitant psoriatic arthritis have contributed in making MTX the drug of choice in managing severe psoriasis. Although the majority of patients achieve remission of disease activity with MTX, a significant proportion may experience mild and transient adverse effects. From time to time, various guidelines on the use of MTX have correctly and adequately stressed the need for strict monitoring of haematological and hepatic adverse events.

The transcription factor known as nuclear factor of kappa light chain enhancer of activated B cells (NF-κB) controls a large number of genes in immune cells in response to inflammation, infection, and other stimuli. Proinflammatory cytokines, chemokines, and growth factors are among the many genes whose transcription is boosted when the NF-κB pathway is activated. These genes are all implicated in the initiation and maintenance of the inflammatory response in psoriatic illness .

The intracellular scaffold protein known as caspase recruitment domain family member 14 (CARD14) rs34367357 is highly abundant in keratinocytes and mediates NF-κB activation by forming a CBM (CARD14-BCL10-MALT1) signaling complex .

Gain-of-function mutations in CARD14 have been demonstrated to increase the development of the CBM complex in keratinocytes, which causes the NF-κB pathway to become hyperactivated. Neutrophils, dendritic cells, and T cells are then drawn in and activated as a result of the transcription of several chemokines (CCL20, CXCL1, and CXCL2), cytokines (IL-36 and IL-19), and antimicrobial peptides. Two key cytokines in the pathophysiology of psoriasis, IL-17 and IL-22, are downstreamly expressed when activated dendritic cells release IL-23 .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* Patients having psoriasis diagnosed clinically and who have a severity grade of moderate to severe, defined as a Psoriasis Area and Severity Index (PASI) score from 5- 10 % of body surface area, and involvement of greater than 10% of the body surface area (BSA) with or without psoriatic arthritis

Exclusion Criteria:

* Patients with other autoimmune conditions (e.g., rheumatoid arthritis, systemic lupus erythematosus).
* Pregnancy and lactation.
* Patients currently undergoing immunosuppressive or systemic therapies.
* Patients with known genetic disorders affect immune system function.
* Patients with liver or kidney impairment.
* Patients with allergy or contraindication to methotrexate.
* Patients with active or uncontrolled infections, including chronic infections like tuberculosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Treatment | 3 Months
  Assessing the Response of psoriasis and psoriatic arthritis to Methotrexate by assessment and complete cutaneous examination to evaluate the clinical type and severity of psoriasis using PASI score

CONTACTS AND LOCATIONS:
Overall Officials: Essam El-Din Abd El-Aziz Mohamed Ahmed Nada, Professor, Study Chair — Dermatology, Venereology and Andrology Sohag university; Eisa Mohammed Hegazy, Professor, Study Director — • Dermatology Venereology & Andrology Faculty of Medicine, South valley University.
Locations (1):
- Qina University hospital, South Valley University Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided